CLINICAL TRIAL: NCT00565370
Title: A Phase I-II Study of Sorafenib (Nexavar®) in Combination With Capecitabine and Cisplatin (XP) in Patients With Advanced Gastric Cancer
Brief Title: Capecitabine and Cisplatin (XP)+Sorafenib in Advanced Gastric Cancer (AGC): Sorafenib+XP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC0701
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Advanced Gastric Cancer
Keywords: Gastric cancer; capecitabine; cisplatin; sorafenib; phase I; phase II
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Cisplatin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): XP+sorafenib
  Interventions: Drug: Capecitabine, Cisplatin, Sorafenib
- B (Placebo Comparator): XP
  Interventions: Drug: Capecitabine, Cisplatin, Sorafenib

INTERVENTIONS:
Drug: Capecitabine, Cisplatin, Sorafenib — Capecitabine ( ) mg/m2 bid D1-D15 Cisplatin 80 mg/m2 D1 Sorafenib ( ) mg bid PO daily every 3 weeks

SUMMARY:
There is strong scientific rationale for exploring the role of sorafenib with capecitabine and cisplatin (XP) in AGC. XP is a new standard of care in AGC and sorafenib is a novel signal transduction inhibitor that prevents tumor cell proliferation and angiogenesis through blockade of the Raf/MEK/ERK pathway at the level of Raf kinase and the receptor tyrosine kinases VEGF-R2 and PDGFR-beta.

ELIGIBILITY:
Inclusion Criteria:

* Having given signed written informed consent
* Unresectable advanced gastric adenocarcinoma, initially diagnosed or recurred
* No history of chemotherapy or radiation
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST)
* Age 18-75 years
* Estimated life expectancy of more than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate bone marrow function (absolute neutrophil count > 1,500/µL, platelets > 100,000/µL, hemoglobin > 8g/dl),
* Adequate kidney function (creatinine clearance > 60 ml/min)
* Adequate liver function (bilirubin < 2.0 mg/dL, transaminases levels < 3 times the upper normal limit [5 times for patients with liver metastasis])

Exclusion Criteria:

* Past or concurrent history of neoplasm other than gastric adenocarcinoma, except for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix uteri
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start
* Presence of central nervous system metastasis
* Obvious peritoneal seeding or bowel obstruction
* Evidence of serious gastrointestinal bleeding
* Peripheral neuropathy (National Cancer Institute Common Terminology Criteria for Adverse Event version 3.0 > Grade I)
* History of significant neurologic or psychiatric disorders
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions
* Known allergy to study drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD, PhD, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- XP Plus Sorafenib: Capecitabine and cisplatin plus sorafenib Level 1 sorafenib 400 mg/d, capecitabine 1,600 mg/m2/d, cisplatin 80 mg/m2 Level 2 sorafenib 800 mg/d, capecitabine 1,600 mg/m2/d, cisplatin 80 mg/m2 Level 3 sorafenib 800 mg/d, capecitabine 2,000 mg/m2/d, cisplatin 80 mg/m2 Level 1A sorafenib 800 mg/d, capecitabine 1,600 mg/m2/d, cisplatin 60 mg/m2
Period: Overall Study
Arm/Group | XP Plus Sorafenib
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled patients were analyzed for analysis.
Groups:
- XP Plus Sorafenib: Capecitabine and cisplatin plus sorafenib
Arm/Group | XP Plus Sorafenib
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 16
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs)
Description: Number of Participants who Experienced Dose Limiting Toxicities (DLTs)
Time Frame: 28weeks
Measure: Number; unit: participants
Arm/Group | XP Plus Sorafenib
Number analyzed (Participants) | 21
participants | 3

2. Primary Outcome: Progression-free Survival
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | XP Plus Sorafenib
Number analyzed (Participants) | 21
Months | 10.0 [7.4 to 13.8]

3. Secondary Outcome: Response Rate
Description: Tumor response was assessed every two cycles by RECIST(v1.0) using the same imaging techniques and methods used at baseline.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar definition that is accurate and appropriate
Time Frame: 6 months
Population: Patients who had measurable lesions were included for the response rates
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XP Plus Sorafenib
Number analyzed (Participants) | 16
percentage of participants | 62.8 [38.8 to 86.2]

4. Secondary Outcome: Overall Survival
Time Frame: 28 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | XP Plus Sorafenib
Number analyzed (Participants) | 21
Months | 14.7 [12.0 to 20.0]

5. Secondary Outcome: Toxicity Profile (According to National Cancer Institute Common Terminology Criteria for Adverse Event Version 3.0)
Description: Number of patients who experienced toxicity from study treatment to evaluate the safety and tolerability of Capecitabine and cisplatin plus sorafenib
Time Frame: 28weeks
Measure: Number; unit: participants
Arm/Group | XP Plus Sorafenib
Number analyzed (Participants) | 21
participants | 21

ADVERSE EVENTS:
Arm/Group | XP Plus Sorafenib
Serious Adverse Events (participants affected / at risk) | 4/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XP Plus Sorafenib (N=21)
Diarrhea (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Deep vein thrombosis (Blood and lymphatic system disorders) | 2
Gastric perforation (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | XP Plus Sorafenib (N=21)
Neutropenia (Blood and lymphatic system disorders) | 14
Leukopenia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Infections and infestations) | 1
Anemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Anorexia (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 13
Stomatitis (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 13
Sensory neuropathy (Nervous system disorders) | 18
Skin rash (Skin and subcutaneous tissue disorders) | 9
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 17
Hypertension (Cardiac disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No